CLINICAL TRIAL: NCT04103125
Title: Open, Non-Comparative Study To Evaluate The Performance And Safety Of The Medical Device JANESSE® (Hyaluronic Acid-Dermal Filler) In The Correction Of Facial Wrinkles
Brief Title: Open, Non-Comparative Study To Evaluate The Performance Of The Medical Device JANESSE®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.A. Istituto Ricerche Applicate S.p.A. (Network)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPIRA/0119/MD
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Wrinkle
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label, non-randomized, single group clinical investigation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Janesse (Other): Janesse® 20 (Cross-linked Hyaluronic Acid) Injection: follow the instruction for use
  Interventions: Device: Janesse® is a sterile, injectable, non-pyrogenic, re-absorbable medical product made of reticulated hyaluronic acid of non-animal origin, produced via bacterial fermentation.

INTERVENTIONS:
Device: Janesse® is a sterile, injectable, non-pyrogenic, re-absorbable medical product made of reticulated hyaluronic acid of non-animal origin, produced via bacterial fermentation. — The subjects will receive at baseline the first IMD by the Investigator in accordance with the CIP

SUMMARY:
The hypothesis of this clinical investigation is that in a population of men and women affected by periocular wrinkles, lip contour wrinkles or deep facial wrinkles, will cross-linked hyaluronic acid (Janesse) significantly decrease the appearance of facial wrinkles, results observed after 4, 8 and 12 weeks.

DETAILED DESCRIPTION:
Janesse®'s action is to increase the volume of dermal-epidermal tissue based on the natural ability of hydrophilic hyaluronic acid molecules to bind to an amount of water many times greater than their weight. This allow to fill the intradermal spaces and integrate the intercellular matrix, conferring turgidity to the tissues. The cross-linking of the hyaluronic acid contained in the product has the effect of more stable and durable filling over time.

The Research Question of the present study is the following: in a population of men and women affected by periocular wrinkles, lip contour wrinkles or deep facial wrinkles, will cross-linked hyaluronic acid (Janesse®) significantly decrease the appearance of nasolabial wrinkles, results observed after 12 weeks?

ELIGIBILITY:
Inclusion Criteria:

1. Men or women with age > 35 and ≤ 65 years.
2. Subjects with nasolabial wrinkles, seeking tissue augmentation treatment and willing to receive HA Filler;
3. Subjects presenting a score of 2 (shallow wrinkles) or 3 (moderate, deep wrinkles) on the Wrinkles Severity Ranking Scale (WSRS);
4. Subjects who agree to discontinue all dermatological treatment and procedures during the study;
5. Subjects willing to provide signed informed consent to clinical investigation participation.
6. Able to communicate adequately with the Investigator and to comply with the requirements for the entire study.

Exclusion Criteria:

1. Subjects who have bleeding disorder in the past or present.
2. Use of aspirin and antiplatelet agents a week prior to treatment
3. Prior or planned use of topical injection to the face (steroid, retinoid: applicable only to drugs, not applicable to cosmetics), within 4 weeks prior to screening or during this study (steroid ointment for therapeutic objectives is allowed for short -term use of ≤14 consecutive days.).
4. Use of immunosuppressive, chemotherapies, or systemic corticosteroids within 12 weeks from screening.
5. History of anaphylaxis or severe complicated allergy symptoms.
6. Clinically significant cardiovascular, digestive, respiratory, endocrine, or central nervous system disorders or previous mental disorders that may significantly affect the study.
7. Hypersensitivity skin reaction to the investigational device based on intradermal test results at screening.
8. Evidence or history of autoimmune disease or compromised immune system.
9. Treatment with anticoagulants, thrombolytics, or platelet inhibitors within 1 week prior to study participation;
10. Prior permanent fillers or fat graft procedures around nasolabial folds.
11. Wrinkle correction procedures (e.g., botulinum toxin A injection, face lift, soft tissue augmentation, medium-depth peel, dermal photorejuvenation, etc.) within 6 months prior to study participation.
12. History of hypersensitivity to local anesthetic of amide type or HA.
13. History of keloid formation or hypertrophic scar on the face.
14. Evidence of active infection on the face.
15. Wound, scar, or skin disorder or infection around nasolabial folds that may affect the efficacy assessment.
16. Pregnant woman, lactating woman, and man or woman of childbearing potential who is planning a pregnancy or is unwilling to use appropriate methods of contraception* during the study, *Methods of contraception: hormonal contraceptive, intrauterine device or intrauterine system, double barrier method (condom with spermicide/diaphragm or cervical cap with spermicide), surgical sterilization (vasectomy, tubal ligation, etc.).
17. As with all dermal filler procedures, the product should not be used in vascular rich areas.
18. Subjects with illness, or other medical condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the study.
19. Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
WSRS score assessed by the Investigator | 12 weeks
  To evaluate the overall safety of the medical device and performance of Janesse® dermal filler in terms of absolute change of WSRS score (Wrinkle Severity Rating Scale) assessed by Investigator at 4, 8 and 12 weeks after the initiation of treatment, compared to Baseline Visit (day 0).
AE, SAE, ADE, SADE incidence | 12 weeks
  AE, SAE, ADE, SADE incidence

SECONDARY OUTCOMES:
WSRS score assessed by the patient | 12 weeks
  To evaluate the performance of the medical device in terms of change of WSRS score assessed by the subject at 4, 8 and 12 weeks compared to Baseline Visit 1 (day 0).
Global Aesthetic Improvement Scale evaluated by the subject | 12 weeks
  Subjects will evaluate their skin appearance change compared to before the treatment, as follows:
  * Very Much Improved (1) = Optimal cosmetic result;
  * Much Improved (2) = Market improvement in appearance but not completely optimal. A touch-up would slightly improve the result;
  * Improved (3) = Obvious improvement in appearance from the initial condition, but a touch-up or re-treatment is indicated;
  * No Change (4) = The appearance is essentially the same as the original condition;
  * Worse (5) = The appearance is worse than the original condition.
Treatment satisfaction questionnaire completed by the subject | 12 weeks
  To assess the subject satisfaction at 4, 8 and 12 weeks, providing their degree of satisfaction with the treatment on a four-point scale (very satisfied, satisfied, moderate or not satisfied).
Investigator Global Assessment of Performance (IGAP) | 12 weeks
  Investigator Global Assessment of Performance (IGAP) Investigator will make photographs at every visit (1, 2, 3, 4 and 5) of the area treated in order to evaluate the performance of the treatment at visit 5 using a 4-point scale: 1= very good performance, 2 = good performance, 3 = moderate performance and 4 = poor performance;taken at each visit.
Investigator Global Assessment of Safety (IGAS) | 12 weeks
  Investigator Global Assessment of Safety (IGAS) will be reported using the 4-point scale: 1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety. IGAS will be evaluated by the Investigator at Final visit (12 weeks), only;
Patient Global Assessment of Safety (PGAS) | 12 weeks
  Patient Global Assessment of Safety (PGAS) will be reported by the subject at the last visit using the 4-point scale: 1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety. PGAS will be evaluated by the patient at Final visit (12 weeks), only.

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Fratila, Principal Investigator — SCM Dr. Rosu
Locations (1):
- SCM Dr. Rosu, Timișoara, Timiș County, Romania

REFERENCES:
- [Background] Fitzgerald R, Graivier MH, Kane M, Lorenc ZP, Vleggaar D, Werschler WP, Kenkel JM. Update on facial aging. Aesthet Surg J. 2010 Jul-Aug;30 Suppl:11S-24S. doi: 10.1177/1090820X10378696. PMID 20844296
- [Background] Kim BW, Moon IJ, Yun WJ, Chung BY, Kim SD, Lee GY, Chang SE. A Randomized, Evaluator-Blinded, Split-Face Comparison Study of the Efficacy and Safety of a Novel Mannitol Containing Monophasic Hyaluronic Acid Dermal Filler for the Treatment of Moderate to Severe Nasolabial Folds. Ann Dermatol. 2016 Jun;28(3):297-303. doi: 10.5021/ad.2016.28.3.297. Epub 2016 May 25. PMID 27274627
- [Background] Few J, Cox SE, Paradkar-Mitragotri D, Murphy DK. A Multicenter, Single-Blind Randomized, Controlled Study of a Volumizing Hyaluronic Acid Filler for Midface Volume Deficit: Patient-Reported Outcomes at 2 Years. Aesthet Surg J. 2015 Jul;35(5):589-99. doi: 10.1093/asj/sjv050. Epub 2015 May 11. PMID 25964628
- [Background] Callan P, Goodman GJ, Carlisle I, Liew S, Muzikants P, Scamp T, Halstead MB, Rogers JD. Efficacy and safety of a hyaluronic acid filler in subjects treated for correction of midface volume deficiency: a 24 month study. Clin Cosmet Investig Dermatol. 2013 Mar 20;6:81-9. doi: 10.2147/CCID.S40581. Print 2013. PMID 23687448
- [Background] Dong J, Gantz M, Goldenberg G. Efficacy and safety of new dermal fillers. Cutis. 2016 Nov;98(5):309-313. PMID 28040813
- [Background] De Boulle K, Heydenrych I. Patient factors influencing dermal filler complications: prevention, assessment, and treatment. Clin Cosmet Investig Dermatol. 2015 Apr 15;8:205-14. doi: 10.2147/CCID.S80446. eCollection 2015. PMID 25926750
- [Background] Rivkin AZ. Volume correction in the aging hand: role of dermal fillers. Clin Cosmet Investig Dermatol. 2016 Aug 30;9:225-32. doi: 10.2147/CCID.S92853. eCollection 2016. PMID 27621659
- [Background] Kuhne U, Esmann J, von Heimburg D, Imhof M, Weissenberger P, Sattler G. Safety and performance of cohesive polydensified matrix hyaluronic acid fillers with lidocaine in the clinical setting - an open-label, multicenter study. Clin Cosmet Investig Dermatol. 2016 Oct 20;9:373-381. doi: 10.2147/CCID.S115256. eCollection 2016. PMID 27799807
- [Background] Lorenc ZP, Bank D, Kane M, Lin X, Smith S. Validation of a four-point photographic scale for the assessment of midface volume loss and/or contour deficiency. Plast Reconstr Surg. 2012 Dec;130(6):1330-1336. doi: 10.1097/PRS.0b013e31826d9fa6. PMID 23190816
- [Background] McCall-Perez F, Stephens TJ, Herndon JH Jr. Efficacy and tolerability of a facial serum for fine lines, wrinkles, and photodamaged skin. J Clin Aesthet Dermatol. 2011 Jul;4(7):51-4. PMID 21779421
- [Background] Rzany B, Cartier H, Kestemont P, Trevidic P, Sattler G, Kerrouche N, Dhuin JC, Ma YM. Full-face rejuvenation using a range of hyaluronic acid fillers: efficacy, safety, and patient satisfaction over 6 months. Dermatol Surg. 2012 Jul;38(7 Pt 2):1153-61. doi: 10.1111/j.1524-4725.2012.02470.x. PMID 22759252
- [Background] Van Dyke S, Hays GP, Caglia AE, Caglia M. Severe Acute Local Reactions to a Hyaluronic Acid-derived Dermal Filler. J Clin Aesthet Dermatol. 2010 May;3(5):32-5. PMID 20725567
- [Background] Funt D, Pavicic T. Dermal fillers in aesthetics: an overview of adverse events and treatment approaches. Plast Surg Nurs. 2015 Jan-Mar;35(1):13-32. doi: 10.1097/PSN.0000000000000087. PMID 25730536
- [Background] Ghooi RB, Bhosale N, Wadhwani R, Divate P, Divate U. Assessment and classification of protocol deviations. Perspect Clin Res. 2016 Jul-Sep;7(3):132-6. doi: 10.4103/2229-3485.184817. PMID 27453830
- [Background] Jiang LI, Stephens TJ, Goodman R. SWIRL, a clinically validated, objective, and quantitative method for facial wrinkle assessment. Skin Res Technol. 2013 Nov;19(4):492-8. doi: 10.1111/srt.12073. Epub 2013 Jun 10. PMID 23750828
- [Background] Stephens TJ, Sigler ML, Herndon JH Jr, Dispensa L, Le Moigne A. A placebo-controlled, double-blind clinical trial to evaluate the efficacy of Imedeen((R)) Time Perfection((R)) for improving the appearance of photodamaged skin. Clin Cosmet Investig Dermatol. 2016 Mar 15;9:63-70. doi: 10.2147/CCID.S98787. eCollection 2016. PMID 27042135